CLINICAL TRIAL: NCT06708338
Title: Impact of Bevel Orientation on Arteriovenous Fistula Puncture in Hemodialysis: A Multicenter Randomized Comparative Study
Brief Title: Impact of Bevel Orientation on Arteriovenous Fistula Puncture in Hemodialysis
Acronym: FAVORI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RIPH2_SOULIER_FAVORI; 2024-A01536-41 (Other: ID-RCB)
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: End-Stage Renal Disease Requiring Haemodialysis
Keywords: arteriovenous fistula; puncture technique; vascular approach
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bevel-up group (Active Comparator): AVF puncture will be performed with the needle bevel facing up for the entire duration of the patient's participation.
  Interventions: Procedure: Needle bevel orientation for arteriovenous fistula puncture
- Bevel-down group (Experimental): AVF puncture will be performed with the needle bevel facing down for the entire duration of the patient's participation
  Interventions: Procedure: Needle bevel orientation for arteriovenous fistula puncture

INTERVENTIONS:
Procedure: Needle bevel orientation for arteriovenous fistula puncture — For the duration of the study (24 months from inclusion), the nurse will puncture the AVF according to the patient's randomization arm.
  Patients will be randomized, according to the minimization technique, in a 1:1 ratio between the following two groups:
  * Bevel-up group
  * Bevel-down group

SUMMARY:
End-stage renal disease (ESRD) is a condition in which the filtration function of the kidneys has deteriorated, necessitating dialysis or transplantation. With an aging population, the number of patients undergoing dialysis for CKD is constantly increasing.

There are different types of dialysis treatment: hemodialysis and peritoneal dialysis.

Hemodialysis involves exchanges between blood and a dialysate (a liquid used to purify blood) via a dialyzer (artificial filter), coordinated by a generator. This method requires a vascular approach, of which there are 3 types: the arteriovenous fistula (AVF), the arteriovenous graft and the central venous catheter.

The AVF remains the vascular access of choice for hemodialysis sessions, and its preservation is an essential objective for patients with CKD.

One of the major challenges for AVFs is to achieve a successful puncture, an act performed around 310 times a year per patient, for dialysis performed three times a week with double needles. This repeated procedure can cause damage to the AVF, leading to complications such as stenosis, thrombosis, aneurysm, superficial infection, hematoma, bleeding, parietal rupture or dissection.

However, there is no official recommendation on the most conservative puncture technique for AVF. In view of the number of patients concerned and the recurrence of puncture, it would seem essential to evaluate the impact of bevel orientation on the occurrence of complications during dialysis by means of a randomized prospective study.

ELIGIBILITY:
Inclusion Criteria:

* male or female with Chronic Kidney Disease
* patient requiring 4-hour hemodialysis sessions, 3 times per week, in a dialysis center
* Native arteriovenous fistula (AVF) (without prosthesis), mature, with no prior puncture, located in the upper limb
* First fistula for a hemodialysis patient
* Expected duration of dialysis ≥ 1 year
* Double-needle dialysis
* Hemodialysis possible on AVF
* Average AVF flow rate between 500 and 2,000 mL/min
* Affiliated with a social security scheme
* Free and informed consent

Exclusion Criteria:

* Auto-dialysis at home
* Puncture using the buttonhole technique
* Patient requiring AVF puncture with a catheter
* Planned transplant within the next 12 months
* Previous AVF creation, except for the fistula of interest
* Patient with a history of cancer within the past 5 years or active cancer
* Patient under court protection or guardianship
* Pregnant and breast-feeding women
* Patient with psychiatric pathologies or cognitive disorders
* Patient follow-up difficult or impossible for geographical or other reasons, at the investigator's discretion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of needle bevel orientation (up versus down) on the occurrence of AVF complications during dialysis sessions over 12 months in patients with ESRD | During dialysis sessions over 12 months, from inclusion
  The primary endpoint is the number of AVF complications over 12 months. Eight AVF complications will be collected (stenosis, thrombosis, aneurysm or aneurysm rupture, pseudoaneurysm, infection, hematoma, bleeding, rupture and/or parietal dissection).

SECONDARY OUTCOMES:
Evaluate, in patients with CKD treated with hemodialysis, the impact of bevel orientation (up versus down) on the occurrence of AVF dysfunction requiring ultrasound during the first 24 months. | For 24 months from inclusion
  Time from insured bipuncture to onset of AVF dysfunction (see complications in primary endpoint) requiring ultrasound over 24 months will be calculated.
Evaluate, in patients with CKD treated with hemodialysis, the impact of bevel orientation (up versus down) on the occurrence of an intervention (surgical or radiointerventional) during the first 24 months | For 24 months from inclusion
  Time from insured bipuncture to onset of AVF dysfunction (see complications in primary endpoint) requiring initial intervention (surgical or radio-interventional) over 24 months will be calculated.
Evaluate, in patients with CKD treated with hemodialysis, the impact of bevel orientation (up versus down) on AVF survival. | For 24 months from inclusion
  The time between the insured bipuncture and the discontinuation of its use over 24 months by the introduction of hemodialysis sessions via a central venous catheter or another AVF will be calculated
Evaluate, in patients with CKD treated with hemodialysis, the impact of bevel orientation (up versus down) on patient discomfort with fistula pain during and between dialysis sessions over 12 months | For 12 months from inclusion
  Patient discomfort score for AVF pain during and between dialysis sessions, assessed using a simple verbal scale with a score ranging from 0 (pain free) to 4 (unbearable pain), at each session over 12 months
Evaluate, in patients with CKD treated with hemodialysis, the impact of bevel orientation (up versus down) on AVF wall thickening at the puncture site at 6, 12 and 24 months. | At 6, 12 and 24 months from inclusion
  Thickening of the AVF wall at the puncture site will be measured in mm by echo-Doppler at 6, 12 and 24 months.
Evaluate caregivers' feedback on the two puncture techniques and any changes in their practice in terms of AVF monitoring. | At Month 12 (if at least 4 patients have been included in the center)
  Feedback from caregivers will be evaluated via a qualitative questionnaire completed every 12 months starting from the fourth patient inclusion in each center. This aims to assess their experience with the two puncture techniques and any impact on their clinical practice.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Hôpital Saint Joseph Saint Luc, Lyon
  - Centre Hospitalier de Moulins-Yzeure, Moulins
  - Ctre Hospitalier Intercommunal Poissy St Germain Site Poissy, Poissy